CLINICAL TRIAL: NCT02827942
Title: Comparison of Dual Amoxicillin/Vonoprazan Therapy and Triple Vonoprazan/Amoxicillin/Clarithromycin or Metronidazole Therapy for H. Pylori Eradication
Brief Title: Comparison of Vonoprazan-based Dual and Triple Therapies for H. Pylori Eradication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamamatsu University (Other)
Responsible Party: Principal Investigator, Takahisa Furuta, Professor, Hamamatsu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R15-006
Record Dates: First submitted 2016-06-12; First posted 2016-07-11 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Gastritis Associated With Helicobacter Pylori
Keywords: pylori
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; BID protein, human; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Intervention Model Description: Comparison of the dual VPZ/AMPC therapy and triple VPZ/AMPC/CAM therapy
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual therapy (Experimental): Patients assigned to this group are treated with dual therapy with vonoprazan 20 mg bid and amoxicillin 500 mg tid for 1 week. The eradication rate attained with this regimen is measured.
  Interventions: Drug: vonoprazan 20 mg bid; Drug: Amoxicillin 500 mg tid
- Triple therapy (Active Comparator): Patients assigned to this group are treated with the triple therapy with vonoprazan 20 mg bid, clarithromycin 200 mg bid and amoxicillin 750 mg bid for 1 week as the first line therapy or the triple therapy with vonoprazan 20 mg bid, metronidazole 250 mg bid and amoxicillin 750 mg bid for 1 week as the second line therapy. The eradication rates attained with these regimens are measured.
  Interventions: Drug: vonoprazan 20 mg bid; Drug: Amoxicillin 750 mg bid; Drug: Clarithromycin 200 mg bid; Drug: Metronidazole 250 mg bid

INTERVENTIONS:
Drug: vonoprazan 20 mg bid — Vonoprazan is potent acid inhibitor. Vonoprazan 20 mg is dosed twice daily for 1 week.
  Other Names: takecab® 20 mg bid
Drug: Amoxicillin 500 mg tid — Amoxicillin is antibiotics. Its bactericidal effect is time-dependent. Then, 500 mg of amoxicillin is dosed three times daily for 1 week.
  Other Names: Sawacillin® 500 mg tid
  Arms: Dual therapy
Drug: Amoxicillin 750 mg bid — Amoxicillin is antibiotics. Its bactericidal effect is time-dependent. However, the standard regimen in Japan, 750 mg of amoxicillin is dosed twice daily with clarithromycin or metronidazole for 1 week. Then, 750 mg of amoxicillin is dosed twice daily.
  Other Names: Sawacillin® 750 mg bid
  Arms: Triple therapy
Drug: Clarithromycin 200 mg bid — Clarithromycin is antibiotics. It is involved in the standard first line regimen in Japan. Then, 200 mg of clarithromycin is dosed twice daily for 1 week.
  Other Names: Claris® 200 mg bid
  Arms: Triple therapy
Drug: Metronidazole 250 mg bid — Metronidazole is antimicrobial agent. It is involved in the standard second line regimen in Japan. Then, 250 mg of metronidazole is dosed twice daily for 1 week.
  Other Names: fragile 250 mg bid
  Arms: Triple therapy

SUMMARY:
Patients infected with H. pylori were randomly assigned to the dual therapy with vonoprazan 20 mg bid and amoxicillin 500 mg tid for 1 week or the triple therapy with vonoprazan 20 mg bid, amoxicillin 750 mg bid and clarithromycin 200 mg or metronidazole 250 mg bid bid for 1 week. Success or failure of eradication was determined by the 13C-urea breath test performed at 1 month after the therapy.

DETAILED DESCRIPTION:
Patients infected with H. pylori were enrolled and invited to the study.

Patients who have never undergone the H. pylori eradication therapy are randomly assigned to the dual therapy with vonoprazan 20 mg bid and amoxicillin 500 mg tid for 1 week or the triple therapy with vonoprazan 20 mg bid, amoxicillin 750 mg bid and clarithromycin 200 mg bid for 1 week.

Patients who have ever failed in the eradication of H. pylori by the triple therapy containing clarithromycin are randomly assigned to the dual therapy with vonoprazan 20 mg bid and amoxicillin 500 mg tid for 1 week or the triple therapy with vonoprazan 20 mg bid, amoxicillin 750 mg bid and metronidazole 250 mg bid for 1 week.

Success or failure of eradication was determined by the 13C-urea breath test performed at 1 month after the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with H. pylori
* Patients who are not allergic to any of drugs used in this study
* Patients who agree to participate to the study patients who are treatment naive for eradication of H. pylori

Exclusion Criteria:

* Patients not infected with H. pylori
* Patients who are allergic to any of drugs used in this study
* Patients who do not agree to participate to the study
* Severe general condition, such as renal insufficiency or liver dysfunction
* History of gastrectomy
* Inability to undergo eradication therapy
* Patients who have ever undergone the eradication therapy for H. pylori infection

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
The success or failure of eradication | 4 to 8 weeks after the end of the eradication therapy
  Success or failure of eradication of H. pylor is to be diagnosed at 4 to 8 weeks after the end of the eradication therapy by13C-urea breath test.

SECONDARY OUTCOMES:
Adverse events | 1 week
  Adverse events related that happen during 1 week-treatments, such as diarrhea, loose stool, abdominal pain, and allergic reaction are checked by interview when patients visit the hospital to undergo the 13C-urea breath test for the diagnosis of success or failure of eradication of H. pylori.

CONTACTS AND LOCATIONS:
Overall Officials: Takahisa Furuta, MD, PhD, Study Chair — Hamamatsu University
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan

IPD SHARING:
Plan to Share IPD: No
The individual data cannot be taken out from the hospital without permission.